CLINICAL TRIAL: NCT07218341
Title: Long-Term Safety of Pirtobrutinib in Participants From Study LOXO-BTK-20020 With BTKi Pretreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study of Pirtobrutinib (LY3527727) in Participants With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27296; J2N-MC-JZ03 (Other: Eli Lilly and Company); J2N-MC-JZNY (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphoma, Small Lymphocytic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib; idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pirtobrutinib (Arm A) (Experimental): Participants receive pirtobrutinib orally
  Interventions: Drug: Pirtobrutinib
- Idelalisib (Arm B) (Experimental): Participants receive idelalisib orally
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally
  Other Names: LY3527727
  Arms: Pirtobrutinib (Arm A)
Drug: Idelalisib — Administered orally
  Arms: Idelalisib (Arm B)

SUMMARY:
This study will evaluate the long-term safety of pirtobrutinib in participants with previously treated chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). The study is open to those who completed J2N-MC-JZNN/LOXO-BTK-20020 (NCT 04666038) for continued access to the study intervention or continued follow-up visits. Treatment will be given every 4 weeks and this study is expected to last about 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Are actively participating in study J2N-MC-JZNN/LOXO-BTK-20020

Exclusion Criteria:

* This is not applicable to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with a Grade 3 or Higher Treatment-emergent Adverse Events (AEs) | Time from First Dose of Study Intervention (Study Day 1) through 30 Days After Last Dose of Study Intervention or Start of New Anticancer Therapy, whichever is Earlier

SECONDARY OUTCOMES:
Overall Survival | Time from Enrollment in the Originator Study until Death from Any Cause (Up to 93 Months)
  Overall survival is defined as the time from randomization in a randomized originator study, or from the first dose in a non-randomized originator study, until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (51):
- United States (9):
  - Mitchell Cancer Institute, Mobile, Alabama
  - Arizona Oncology Associates, P.C. - HOPE, Tucson, Arizona
  - Cancer Specialists, LLC, Jacksonville, Florida
  - University of Maryland, Baltimore, Maryland
  - Minnesota Oncology Hematology, P.A., Coon Rapids, Minnesota
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Texas Oncology - Paris, Fort Worth, Texas
  - US Oncology - Texas Oncology, Kyle, Texas
- Australia (2):
  - Liverpool Hospital, Liverpool
  - The Alfred Hospital, Melbourne
- LKH - Universitätsklinikum der PMU Salzburg, Salzburg, Austria
- AZ Delta, Roeselare, Belgium
- Princess Margaret Cancer Centre - University Health Network, Toronto, Canada
- China (11):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Sun Yat-sen University Cancer Center, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Gansu Provincial Cancer Hospital, Lanzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
- University Hospital Center Zagreb, Zagreb, Croatia
- France (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Kralove
  - Centre Henri Becquerel, Rouen
- Hungary (2):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem, Debrecen
- Ireland (2):
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
- Italy (9):
  - Azienda Ospedaliero - Universitaria Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Presidio Ospedaliero Papardo, Messina
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Azienda Ospedaliera S. Maria Di Terni, Terni
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma, Verona
- Tokai University Hospital, Isehara, Japan
- Poland (4):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny im.ks.B.Markiewicza, Brzozów
  - Szpital Uniwersytecki Nr 2 im. dr J. Biziela w Bydgoszczy, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Instytut Hermatologii I Transfuzjologii, Warsaw
- Spain (2):
  - Hospital Universitario Marques De Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (3):
  - Castle Hill Hospital, Hull
  - St James's University Hospital, Leeds
  - GenesisCare, Newmarket

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement
URL: http://vivli.org/